CLINICAL TRIAL: NCT00000521
Title: Sodium-Potassium Blood Pressure Trial in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 40; R01HL034659 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, potassium-supplemented

SUMMARY:
To examine the effects of nutritional intervention on the rate of rise of blood pressure in late childhood and early adolescence.

DETAILED DESCRIPTION:
BACKGROUND:

Since 1970, children and adolescents with hypertension have been detected with increasing frequency. Many of them were thought to have primary or essential hypertension and it remained unclear how they should be managed. Additionally, since tracking of blood pressure occurred even in early life, it was believed that youngsters with blood pressures persistently in the upper deciles for age were at increased risk for later hypertension. No clinical trials had been performed in this age group to examine the effects of non-pharmacologic or drug therapy in lowering blood pressure. The trial was one of the first attempts to examine the effects of a nutritional intervention on the rate of rise of blood pressure in late childhood and early adolescence.

DESIGN NARRATIVE:

Randomized, partial-blind. After 19,542 fifth to eighth grade students were screened, 210 (105 boys and 105 girls) from the upper 15 percentiles of blood pressure distribution were randomly assigned to one of three groups: low sodium diet (70 mmol sodium intake per day), potassium chloride supplementation (normal diet plus 1 mmol/kg potassium chloride per day), and placebo (normal diet plus placebo capsule). Capsules for the potassium chloride and placebo groups were administered in a double blind protocol. Blood pressure was measured every three months for three years. The effect of the intervention was determined by comparing the rate of rise (slope) of blood pressure among the groups using a random-coefficient growth curve model.

ELIGIBILITY:
Children in grades 5 through 8 whose systolic blood pressure was greater than or equal to 120 mm Hg on two visits.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 1985-08; Primary Completion 1990-07 (Actual); Study Completion 1990-12 (Actual)

REFERENCES:
- [Background] Gomez-Marin O, Prineas RJ, Sinaiko AR. The Sodium-Potassium Blood Pressure Trial in Children. Design, recruitment, and randomization: the children and adolescent blood pressure program. Control Clin Trials. 1991 Jun;12(3):408-23. doi: 10.1016/0197-2456(91)90020-m. PMID 1651211
- [Background] Sinaiko AR, Gomez-Marin O, Prineas RJ. Effect of low sodium diet or potassium supplementation on adolescent blood pressure. Hypertension. 1993 Jun;21(6 Pt 2):989-94. doi: 10.1161/01.hyp.21.6.989. PMID 8505112